CLINICAL TRIAL: NCT00945529
Title: The Effects of Inhaled Nitric Oxide on Patient Morbidity and Length of Hospital Stay Following Fontan Operation
Brief Title: The Effects of Inhaled Nitric Oxide After Fontan Operation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ellen Spurrier (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Ellen Spurrier, Director of Cardiac Anesthesiology, Nemours Children's Clinic
Organization: Nemours Children's Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPURE1
Record Dates: First submitted 2009-05-28; First posted 2009-07-24 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Defect
Keywords: Fontan
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Intervention/ historical control group (No Intervention): historical controls group of patients who did not receive iNO.
- Intervention (Experimental): Prospective group who received iNO.
  Interventions: Drug: inhaled nitric oxide (iNO)

INTERVENTIONS:
Drug: inhaled nitric oxide (iNO) — Inhaled nitric oxide 40ppm for 48 hours followed by a 6-hour wean.
  Other Names: Inomax
  Arms: Intervention

SUMMARY:
Pleural effusions continue to be a post-operative complication seen after Fontan operation. This study will examine the use inhaled nitric oxide (iNO) given for 54 hours after Fontan operation to improve fluid balance. The study hypothesis is that inhaled nitric oxide after Fontan operation will improve fluid balance, thus decreasing the incidence of pleural effusions and shortening hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients
* Undergoing Fontan operation at the Nemours Cardiac Center at A. I. duPont Hospital for Children
* Written parental permission to participate in this research study

Exclusion Criteria:

* Any condition which the PI feels will interfere with the patient's safe and effective participation

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Spurrier, MD, Principal Investigator — Nemours Children's Clinic - A. I. duPont Hospital for Children
Locations (1):
- A. I. duPont Hospital for Children/Nemours Cardiac Center, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective participant recruitment took place between February 2008 and December 2010 at the Nemours Cardiac Center at A. I. duPont hospital for Children.
Groups:
- Intervention: Prospective group who received iNO.
  inhaled nitric oxide: Inhaled nitric oxide 40ppm for 48 hours followed by a 6-hour wean.
Period: Overall Study
Arm/Group | No Intervention/ Historical Control Group | Intervention
Started (Data collection only - waiver of consent) | 23 (Historical controls consisted of patients prior to February 2008 who did not receive iNO.) | 21
Completed | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Prospective intervention group - consent obtained prior to research activity Historical control group - data collection only - waiver of consent
Groups:
- No Intervention/ Historical Control Group: historical controls group of patients who did not receive iNO / data collected under waiver of consent
- Intervention: Prospective group who received iNO / Consent obtained
  inhaled nitric oxide: Inhaled nitric oxide 40ppm for 48 hours followed by a 6-hour wean.
- Total: Total of all reporting groups
Arm/Group | No Intervention/ Historical Control Group | Intervention | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Full Range); unit: months] | 18.5 [12 to 36] | 21.0 [14 to 36] | 19.7 [12 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 18 | 13 | 31
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay Following Fontan
Time Frame: until hospital discharge
Measure: Mean (Full Range); unit: days
Arm/Group | No Intervention/ Historical Control Group | Intervention
Number analyzed (Participants) | 23 | 21
days | 11.2 [4 to 60] | 11 [4.5 to 31]

2. Secondary Outcome: Percent of Patients With Significant Pleural Fluid Collections That Required Thoracostomy Drainage
Description: Percent of patients with significant pleural fluid collections that required thoracostomy drainage
Time Frame: 2 weeks
Measure: Number; unit: percentage
Arm/Group | No Intervention/ Historical Control Group | Intervention
Number analyzed (Participants) | 23 | 21
percentage | 43.5 | 33.4

ADVERSE EVENTS:
Arm/Group | No Intervention/ Historical Control Group | Intervention
Serious Adverse Events (participants affected / at risk) | 8/23 | 5/21
Other Adverse Events (participants affected / at risk) | 7/23 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention/ Historical Control Group (N=23) | Intervention (N=21)
prolonged hospital stay due to infection (Infections and infestations) | 5 (5) | 2 (2)
Prolonged hospital stay due to feeding issue (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — feeding intolerance with hyponatremia
Prolonged hospital stay due to atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Prolonged hospital stay due to pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Prolonged hospital stay due to seizures (Nervous system disorders) | 1 (1) | 0 (0)
Prolonged hospital stay due to SVT (Cardiac disorders) | 1 (1) | 0 (0)
Reoperation (Surgical and medical procedures) | 0 (0) | 1 (1) — Superior Vena Cava (SVC) stenosis and large lateral tunnel fenestration after Fontan which required reoperation.
Prolonged hospital stay due to sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention/ Historical Control Group (N=23) | Intervention (N=21)
Pleural effusion requiring drainage (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No